CLINICAL TRIAL: NCT02414178
Title: F 18 T807 Tau PET Imaging in Dominantly Inherited Alzheimer's Network (IND 123119, Protocol D
Brief Title: F 18 T807 Tau PET Imaging in Dominantly Inherited Alzheimer's Network (DIAN Project)
Acronym: AV ADAD
Status: Enrolling by invitation | Type: Observational
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Principal Investigator, Tammie L. S. Benzinger, MD, PhD, Professor of Radiology & Neurological Surger, Washington University School of Medicine
Other Study IDs: IND 123119 Protocol D
Record Dates: First submitted 2015-04-07; First posted 2015-04-10 (Estimated); Last update posted 2025-06-10 (Actual); Status verified 2025-06

CONDITIONS: Alzheimer Disease
Keywords: Dementia; Brain Diseases; Central Nervous System Diseases; Mild Cognitive Impairment; nervous system diseases; Neurodegenerative Disease
MeSH Terms: conditions — Alzheimer Disease; Dementia; Brain Diseases; Central Nervous System Diseases; Cognitive Dysfunction; Nervous System Diseases; Neurodegenerative Diseases | interventions — 7-(6-fluoropyridin-3-yl)-5H-pyrido(4,3-b)indole

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Experimental F 18 T807
  Interventions: Drug: F 18 T807

INTERVENTIONS:
Drug: F 18 T807 — Participants will receive a single intravenous bolus injection of approximately 6.5-10mCi (240-370MBq) of F 18 T807. For those who cannot tolerate the full exam, participants will receive single intravenous bolus injection of approximately 6.5-10mCi (240-370MBq) of F 18 T807.
  Other Names: 18F-AV-1451

SUMMARY:
The purpose of this research study is to evaluate a new radioactive compound used in positron emission tomography (PET) scans in identifying tau tangles (a certain protein that might be associated with Dominantly Inherited Alzheimer's Disease) in the brain, and if the amount of tau tangles in the brain has a relationship to cognitive status.

This study involves a PET scans using the radioactive compound, F 18 T807 for measurement of tau deposition. This radioactive compound is not approved by the United States Food and Drug Administration (FDA). An MRI may also be conducted.

DETAILED DESCRIPTION:
The investigators hypothesize that in vivo tau imaging will ultimately:

* Demonstrate the presence of tau fibrils in the brain during the pre-symptomatic stages of cognitive decline, prior to cerebral atrophy, hypometabolism (as measured by 18F-FDG PET imaging), and dementia.
* Demonstrate that the phenoconversion from cognitively normal (CN) status to early stages of cognitive impairment will be closely correlated with neocortical F 18 T807 uptake and that amyloid positive CN individuals who are positive for F 18 T807 will demonstrate conversion to early dementia.
* Correlate closely with the appearance of CSF markers of tau, including tau, p-tau, and VILIP-1.
* Co-localize with specific cognitive deficits (i.e. patients with tau deposition in the left lateral temporal lobe will have primarily language deficits).
* Predict the onset of dementia more accurately than existing biomarkers.

ELIGIBILITY:
Inclusion Criteria:

1. Participants have met all eligibility criteria for enrollment into the "Dominantly Inherited Alzheimer's Network (DIAN) Performance Site" (IRB ID: 201109187) or the DIAN Extended Registry (EXR)
2. Male or female participants, at least 18 years of age
3. Cognitively normal, or with mild dementia, as assessed clinically
4. Participant is able and willing to undergo testing (MRI or CT, PET, radioactive tracer injection; for those unable to undergo an MRI, CT will be used to generate regions-of-interest).
5. Pre-menopausal women will undergo a urine pregnancy test within 24 hours of drug administration. Only negative pregnancy test result would allow the drug administration to proceed.

Exclusion Criteria:

1. Has any condition that, in the Investigator's opinion, could increase risk to the participant, limit the participant's ability to tolerate the experimental procedures, or interfere with the collection/analysis of the data (for example, participants with severe chronic back pain might not be able to lie still during the scanning procedures).
2. Is deemed likely unable to perform the imaging procedures for any reason.
3. Has a high risk for Torsades de Pointes or is taking medications known to prolong QT interval.
4. Has hypersensitivity to F 18 T807 or any of its excipients.
5. Contraindications to PET, PET-CT or MR (e.g. electronic medical devices, inability to lie still for long periods) that make it unsafe for the individual to participate.
6. Severe claustrophobia.
7. Women who are currently pregnant or breast-feeding, and women who do not agree to use reliable contraception, or to refrain from sexcual activity for 24 hours following administration of the flortaucipir injection will be excluded from the study.
8. Other than DIAN study, currently participating in any research study and receiving an active study medication for Alzheimer's Disearse, an investigational drug, device, imaging, or placebo within the past 30 days before screening, and throughout this clinical trial up to 2-weeks past any study-related procedures.
9. Other than DIAN study, current or recent (within 12 months prior to screening) participation in research studies involving radioactive agents such that the total research-related radiation dose to the participant in any given year would exceed the limits set forth in the US Code of Federal Regulations (CFR) Title 21 Section 361.1. http://www.accessdata.fda.gov/scripts/cdrh/cfdocs/cfcfr/CFRSearch.cfm?FR=361.1. It is the responsibility of each site to confirm the date of the most recent PET scan and to work within the guidelines of the local Radioactive Drug Research Committee (RDRC) regarding the imaging interval.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants are enrolled in the "Dominantly Inherited Alzheimer's Network (DIAN) Performance Site" (IRB ID: 201109187) or the DIAN Extended Registry (EXR)
Sampling Method: Non-Probability Sample
Enrollment: 130 (Estimated)
Dates: Start 2021-03-01 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
F 18 T807 Standard Uptake Value Ratios (SUVR) will be correlated with other imaging modalities (MRI, PET amyloid imaging) and cognitive performance. | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Tammie Benzinger, MD, PhD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States